CLINICAL TRIAL: NCT06502327
Title: Comparison of Visual Instructions for Inserting a Laryngeal Mask in a Neonatal Mannequin [Comparación de Instructivos Para inserción de máscara laríngea en maniquí Neonatal].
Brief Title: Comparison of Visual Instructions for Inserting a Laryngeal Mask in a Neonatal Mannequin.
Acronym: Neo-LMi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of San Marcos, Peru (Other)
Responsible Party: Principal Investigator, Carlos A. Delgado, Associate Research Professor, National University of San Marcos, Peru
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A24011761
Record Dates: First submitted 2024-07-01; First posted 2024-07-16 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Cardiopulmonary Resuscitation; Newborn Asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instructions A (Experimental): The "Instructions A" is a four-step, coloured illustrated brochure with images of newborn mannequins and supplies for laryngeal mask insertion.
  Interventions: Other: Instructions A
- Instructions B (Active Comparator): The "Instructions B" is a six-step, black-and-white illustrated brochure with images of adults and supplies for laryngeal mask airway insertion.
  Interventions: Other: Instructions B

INTERVENTIONS:
Other: Instructions A — "Instructions A" are printed visual instructions for health students for inserting a laryngeal mask into neonatal mannequins.
  Arms: Instructions A
Other: Instructions B — "Instructions B" are printed visual instructions for health students for inserting a laryngeal mask into neonatal mannequins.
  Arms: Instructions B

SUMMARY:
This research project compares the effectiveness of two visual instructions for inserting laryngeal masks. Researchers will assess the procedure performed by undergraduate health students on neonatal mannequins. The student's performance will be evaluated by assessing the results, timing and sequence recorded in videos during the simulation. An Ethical Committee reviewed and approved the protocol.

DETAILED DESCRIPTION:
This research project compares the effectiveness of two visual instructions for inserting laryngeal masks. Researchers will assess the procedure performed by undergraduate health students on neonatal mannequins. The students will participate voluntarily after signing an informed consent. The participating students will be randomly assigned to one of the two groups, each receiving a different visual instruction. The student's performance will be evaluated by assessing the results, timing and sequence recorded in videos during the simulation. An Ethical Committee reviewed and approved the protocol. The Universidad Nacional Mayor de San Marcos funded the investigation through the 2024 grant contest for Research Groups.

The project aims to provide evidence of the advantages of visual instructional methods for inserting laryngeal masks, which contribute to advancing knowledge in medical training and neonatal procedures. The results are expected to inform the selection of more effective educational materials, thus improving student preparation and neonatal care. This research has the potential to bridge the gap between academic theory and clinical practice, benefiting both society and scientific development in neonatal medicine.

ELIGIBILITY:
Inclusion Criteria:

* Students, Health Occupations
* In the last year of studies at the University of San Marcos or any other similar University, and having basic knowledge of neonatal procedures.

Exclusion Criteria:

* Student not registered or withdrawn from courses
* Not having signed the informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants achieving effective ventilation. | Through study completion, an average of six months.
  Effective ventilation with a manual resuscitator involves the inflow of air into the mannequin's lungs through the laryngeal mask and raising the thorax.

SECONDARY OUTCOMES:
Timing measures in the procedure. | From the start of the review of instructions to the verification of chest expansion or failure to achieve chest expansion with at least three ventilation, whichever came first, assessed up to 10 minutes.
  The time, as recorded in a video, captures the entire process, including the required time to review instructions, the moment of laryngeal mask placement, the start of positive pressure ventilation, and the verification of the mannequin's chest expansion with ventilation.
Number of participants achieving a correct sequence. | Through study completion, an average of six months.
  The correct sequence, involves the initial use of a syringe to extract air, the placement of the laryngeal mask, and the final use of the syringe to inject air, before ventilation with a manual resuscitator.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Delgado, MD, PhD, Principal Investigator — National University of San Marcos, Peru
Locations (1):
- Faculty of Medicine. Simulation Center., Lima, Peru